CLINICAL TRIAL: NCT07218588
Title: Sanctuary Farm Prescription in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Carissa Baker-Smith, Director of Research, Nemours Cardiac Center; Director of Preventive Pediatric Cardiology, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000466; ITPR2025333 (Other: Nemours ITP Number)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity &Amp; Overweight; Adolescence
Keywords: adolescence; obesity; overweight; diet
MeSH Terms: conditions — Obesity; Overweight | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Produce prescription (Experimental): weekly produce pickup
  Interventions: Other: dietary / produce

INTERVENTIONS:
Other: dietary / produce — 8-week produce prescription pickup

SUMMARY:
The goal of this research study is to learn if an 8-week produce prescription program (in partnership with a local urban farm) can increase fruit and vegetable consumption in overweight teens and improve their blood pressure and weight. The main questions are:

* Is a produce prescription program in overweight teens feasible?
* Will a produce prescription with educational videos increase weekly fruit and vegetable intake?
* Will a produce prescription with educational videos improve blood pressure and weight for height?

Researchers will compare the teens' fruit and vegetable intake, blood pressure and weight for height before and after the produce prescription. Researchers will also see how feasible it is by measuring the number of produce prescriptions are picked up by the families and how many educational videos are viewed.

Participants will:

* complete questionnaires related to their diet and nutrition
* measure their blood pressure and weight at the beginning and end of the study
* obtain weekly produce prescriptions

DETAILED DESCRIPTION:
The overall objectives of this study are to (1) assess the feasibility of produce-prescription in partnership with a local urban farm (Sanctuary Farm) and to (2) determine if an 8-week produce prescription combined with four 20-minute educational videos improves weekly fruit and vegetable intake and improves BMI and BP in adolescents with dysfunctional adiposity. We hypothesize that implementing a produce prescription program in partnership with a local urban farm is feasible and can potentially overcome barriers to healthy eating. Our team of clinicians and health educators has extensive experience leading dietary intervention studies and community-engaged, patient-centered research.

ELIGIBILITY:
Inclusion

1. Patients seen at Nemours TJU Primary Care Clinic
2. Ages 12-17 years at enrollment
3. BMI > or = 85th percentile
4. English Speaking
5. Willing to provide parental permission and ability to provide child assent for the study

Exclusion

1. Children with neurocognitive delays that would limit participation or ability to assent
2. Use of G-tube/J-tube
3. Food allergies that in the opinion of the investigators would interfere with ability to participate.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent produce pickups completed | 8 weeks
  Percent of produce pickups completed
Percent of videos viewed | 8 weeks
  Percent of educational videos viewed

SECONDARY OUTCOMES:
Change in Blood Pressure | 8 weeks
  Change in blood pressure from baseline
Change in BMI | 8 weeks
  Change in BMI from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Carissa Baker-Smith, MD, MPH, MS, Principal Investigator — Nemours Children's Hospital
Locations (3):
- United States (3):
  - Nemours Children's Hospital, DE, Wilmington, Delaware
  - Nemours Children's Health, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No